CLINICAL TRIAL: NCT05355298
Title: A Phase 1b/2a, Multicentre, Open Label Study of the Pharmacokinetics, Safety and Efficacy of AMP945 in Combination with Nab-paclitaxel and Gemcitabine in Pancreatic Cancer Patients
Brief Title: ACCENT: AMP945 in Combination with Nab-paclitaxel and Gemcitabine for Treatment of Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amplia Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMP945-PC-201
Record Dates: First submitted 2022-04-07; First posted 2022-05-02 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer; PDAC; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm study but 2 parts;
  * Part A is dose escalation
  * Part B is open label single dose level
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AMP945 (Experimental): Part A: AMP945 administered in dose escalating cohorts Part B: AMP945 recommended phase 2 dose
  Interventions: Drug: AMP945 ascending doses; Drug: AMP945 RP2D

INTERVENTIONS:
Drug: AMP945 ascending doses — Part A is a phase 1b dose-escalation design that will enrol at least 3 participants in each of 4 dose-level cohorts, to determine the RP2D of AMP945 to be explored in Part B. Dose escalation decisions will be made using a standard 3+3 dose-escalation phase 1 oncology study design.
Drug: AMP945 RP2D — Part B will determine the efficacy of the AMP945 priming regimen at the recommended phase 2 dose (RP2D) determined in Part A.

SUMMARY:
This is a multicentre, open label, two-part study to determine whether the focal adhesion kinase (FAK) inhibitor AMP945, when given prior to dosing with gemcitabine and nab-paclitaxel, improves response to therapy in first-line patients with unresectable or metastatic pancreatic cancer.

Part A is a phase 1b dose-escalation design that will enrol at least 3 participants in each of 4 dose-level cohorts, to determine the RP2D of AMP945 to be explored in Part B.

Part B will determine the efficacy of the AMP945 regimen at the RP2D, and will be run as a Simon Two-stage design; Stage 1 will enrol 26 participants. If ≤5 of the 26 participants show an objective response, then recruitment will be paused and a detailed analysis of futility will be performed. If the study is deemed futile, recruitment will cease. If the study is determined to be not futile or >5 of the 26 participants show an objective response, recruitment will continue, and an additional 24 participants will be enrolled in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study procedures and agree to adhere to all protocol requirements.
2. Aged at least 18 years at the time of consent.
3. Confirmed histological or cytological diagnosis of advanced pancreatic adenocarcinoma that is:

   Part A: metastatic or not surgically resectable.

   Part B: metastatic, with initial diagnosis of metastatic disease ≤6 weeks prior to Baseline.
4. Has measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
5. Eligible for treatment with nab-paclitaxel and gemcitabine as standard of care therapy.
6. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1, sustained on two separate assessments: the first at least 2 weeks prior to the 1st dose of AMP945 and the 2nd within 72 hours prior to the 1st dose of AMP945. Participants not maintaining an ECOG Performance Score of 0-1 at the second assessment will be excluded from participation.
7. Has a life expectancy of >3 months.
8. Adequate organ function, as defined by the laboratory results below (samples must be obtained ≤14 days prior to study drug administration):

   a) Haematology:

   (i) Absolute neutrophil count (ANC) ≥1.5 × 109/L;

   (ii) Platelet count ≥100,000/mm3 (100 × 109/L);

   (iii) Haemoglobin (Hgb) ≥9 g/dL.

   b) Serum chemistry:

   (i) Aspartate transaminase (AST) (SGOT), ALT (SGPT) ≤2.5 × upper limit of normal range (ULN), unless liver metastases are clearly present, then ≤5 × ULN is allowed;

   (ii) Total bilirubin ≤ULN;

   (iii) Creatinine <1.5 x upper limit of normal (ULN) or estimated glomerular filtration rate (eGFR) >60 mL/min/1.73m2 (calculated using the Cockcroft-Gault equation).

   c) No clinically significant abnormalities in coagulation results.

   d) No clinically significant abnormalities in urinalysis results.
9. Agree to use contraception according to protocol

Exclusion Criteria:

1. Pregnant or breast-feeding, or plans to become pregnant during the study.
2. Has received any investigational medicinal product (IMP) within 30 days or 5 half-lives (whichever is longer) prior to Day -8.
3. Known brain metastases, unless previously treated and well-controlled for at least 3 months (defined as clinically stable, no oedema, no steroids and stable in 2 scans at least 4 weeks apart).
4. Gastrointestinal condition that could interfere with the swallowing or absorption of study medication.
5. Part A: Has received prior systemic treatments for pancreatic cancer, except those given in the adjuvant setting, and with recurrence more than 6 months after completion of curative/adjuvant treatment.
6. Part B: Has received no previous radiotherapy, surgery, chemotherapy, or investigational therapy for the treatment of metastatic disease. Prior treatment with 5-FU or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present. Participants having received cytotoxic doses of gemcitabine or any other chemotherapy in the adjuvant setting are not eligible for this study.
7. History of malignancy other than in situ cancer or basal or squamous cell skin cancer in the last 5 years.
8. Major surgery, other than diagnostic surgery (i.e., surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day -8.
9. Known human immunodeficiency virus (HIV) and/or history of Hepatitis B or C infections or known to be positive for Hepatitis B surface antigen (HBsAg) or Hepatitis C Antibody.
10. Known history of myocardial infarction, coronary stenting, stroke, or cerebrovascular accident within 6 months prior to the first dose of study drug.
11. Focal palliative radiotherapy (e.g., to a bony metastasis) within the 14 days prior to Run-in, or more extensive radiotherapy within 28 days prior to Run-in.
12. History of chronic leukemias (e.g., chronic lymphocytic leukemia).
13. History of interstitial lung disease, history of slowly progressive dyspnoea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.
14. History of connective tissue disorders (e.g., lupus, scleroderma, arteritis nodosa).
15. Clinical signs of active infection and/or a temperature of > 38.0°C at the time of Screening or Baseline. Study entry may be deferred at the discretion of the Principal Investigator (PI).
16. Currently using warfarin.
17. Administration of a live virus vaccine in the 4 weeks prior to Day -8 or plans to receive a live virus vaccine during the study.
18. Clinically significant allergies to AMP945, nab-paclitaxel or gemcitabine (or any of their excipients), including hypersensitivity reactions to human albumin, that are not likely to be well controlled with premedication or other supportive measures.
19. Exhibiting any of the conditions or events outlined in the Contraindications or Special Warnings and Precautions sections of the nab-paclitaxel and/or gemcitabine package inserts.
20. Peripheral neuropathy > Grade 1.
21. Corrected QT interval using Fridericia's correction (QTcF) > 460 ms for males and >480 ms for females.
22. Any clinically relevant medical, social, or psychiatric conditions, or any finding during Screening, which in the Investigator's opinion may put the participant at unacceptable risk or interfere with the study objectives.
23. Prior treatment with AMP945.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) from Baseline to End of Study | From first dose of study drug to end of study, an expected average of 6 months
  TEAEs during study treatment and follow up periods
Part A: Determination of RP2D | After Cycle 1 (28 days) for each Part A cohort
  The RP2D of AMP945 will be determined based on either the maximum tolerated dose or maximum pharmacodynamic effect, which ever is reached first
Part B: efficacy of AMP945 | Imaging every 56 days per participant, with an expected average duration of 6 months
  Overall response rate based on RECIST 1.1

SECONDARY OUTCOMES:
Part A: efficacy of AMP945 | Imaging every 56 days per participant, with an expected average duration of 6 months
  Overall response rate based on RECIST 1.1
AMP945 levels in plasma | Days -8, -7, 1, 3, 4, 8 and 10
  Measurement of maximum concentration (cmax) of AMP945
AMP945 levels in plasma | Days -8, -7, 1, 3, 4, 8 and 10
  Measurement of time to cmax (tmax)
AMP945 levels in plasma | Days -8, -7, 1, 3, 4, 8 and 10
  Measurement of clearance (CL)

OTHER OUTCOMES:
Overall response | Imaging every 56 days per participant, with an expected average duration of 6 months
  Overall response, based on RECIST, by imaging timepoint
Duration of response (DOR) | Imaging every 56 days per participant, with an expected average duration of 6 months
  DOR based on RECIST defined as the time from the date of the first confirmed response to the date of progression or death
Overall survival (OS) | Imaging every 56 days per participant, with an expected average duration of 6 months
  OS of participants, defined as time from first dose until death from any cause
Progression free survival (PFS) | Imaging every 56 days per participant, with an expected average duration of 6 months
  PFS of participants, defined as time from first dose to date of first observed progression, based on RECIST, or death from any cause (whichever comes first)
Time to progression | Imaging every 56 days per participant, with an expected average duration of 6 months
  Time to progression, defined as time from first dosing to date of first observed progression, based on RECIST
Clinical benefit rate (CBR) | Imaging every 56 days per participant, with an expected average duration of 6 months
  CBR defined as complete response (CR) + partial response (PR) + stable disease
Effects on tumor antigens | Every 28 days per participant, with an expected average duration of 6 months
  Changes in levels of tumour antigens (serum CA19-9) at the end of each treatment cycle compared to baseline
Effects on biomarkers | Every 28 days per participant, with an expected average duration of 6 months
  Change in levels of other relevant blood biomarkers including p-FAK, PRO-C3, PRO-C6, PRO-C11, C3M, C6M, and C4G

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (8):
  - GenesisCare, St Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Gallipolli Medical Research Foundation, Greenslopes, Queensland
  - Epworth Healthcare, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Western Health, St Albans, Victoria
- South Korea (5):
  - National Cancer Centre, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Severence Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung Medical Centre, Seoul

IPD SHARING:
Plan to Share IPD: No